CLINICAL TRIAL: NCT05948072
Title: Pre-and Post-operative Cetuximab Plus mFOLFOX6 Versus mFOLFOX6 Alone in RAS/BRAF Wild Type Patients With High-Risk Resectable Colorectal Liver Metastases
Brief Title: Cetuximab+mFOLFOX6 VS. mFOLFOX6 Alone in RAS/BRAF Wild Type Patients With High-Risk Resectable CRLM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director of the Department of Colorectal Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEO-HR-CRLM
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mFOLFOX6 + Cetuximab (Experimental): Cetuximab + mFOLFOX6: Cetuximab (500mg/m2 IV ) will be given. Oxaliplatin (85 mg/m2 IV over 2 h on day 1), Leucovorin calcium (350 mg/m2 IV over 2 h on day 1) plus a bolus of 5FU (400 mg/m2) followed by a 46h-48h IV infusion of 5FU 2400 mg/m2 will be repeated for every 2 weeks. The regimens repeat every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: mFOLFOX6 + Cetuximab
- mFOLFOX6 (Active Comparator): mFOLFOX6: Oxaliplatin (85 mg/m2 IV over 2 h on day 1), Leucovorin calcium (350 mg/m2 IV over 2 h on day 1) plus a bolus of 5FU (400 mg/m2) followed by a 46h-48h IV infusion of 5FU 2400 mg/m2 will be repeated for every 2 weeks. The regimens repeat every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: mFOLFOX 6

INTERVENTIONS:
Drug: mFOLFOX6 + Cetuximab — Cetuximab + mFOLFOX6: Cetuximab (500mg/m2 IV ) will be given. Oxaliplatin (85 mg/m2 IV over 2 h on day 1), Leucovorin calcium (350 mg/m2 IV over 2 h on day 1) plus a bolus of 5FU (400 mg/m2) followed by a 46h-48h IV infusion of 5FU 2400 mg/m2 will be repeated for every 2 weeks. The regimens repeat every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Arms: mFOLFOX6 + Cetuximab
Drug: mFOLFOX 6 — mFOLFOX6: Oxaliplatin (85 mg/m2 IV over 2 h on day 1), Leucovorin calcium (350 mg/m2 IV over 2 h on day 1) plus a bolus of 5FU (400 mg/m2) followed by a 46h-48h IV infusion of 5FU 2400 mg/m2 will be repeated for every 2 weeks. The regimens repeat every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Arms: mFOLFOX6

SUMMARY:
For patients with initially resectable colorectal cancer liver metastases who have high-risk factors, neoadjuvant therapy is currently considered a consensus approach. However, there is ongoing debate regarding the optimal treatment strategy. Our study aims to investigate whether the addition of cetuximab to neoadjuvant chemotherapy improves outcomes compared to neoadjuvant chemotherapy alone. The objective of this phase III clinical trial is to determine whether the combination of cetuximab and mFOLFOX6 chemotherapy is superior to neoadjuvant mFOLFOX6 chemotherapy alone for patients with initially resectable colorectal cancer liver metastases who have wild-type RAS/BRAF and high-risk factors.

DETAILED DESCRIPTION:
Primary

• To determine whether the addition of cetuximab to neoadjuvant mFOLFOX6 chemotherapy results in improved event-free survival when compared with neoadjuvant mFOLFOX6 chemotherapy alone in patients with high-risk & RAS/BRAF-wild-type & resectable colorectal liver metastases.

Secondary

* To evaluate the overall survival of patients treated with these regimens.
* To evaluate the quality of life of patients treated with these regimens.
* To evaluate the preoperative remission rate, safety, surgical complications, actual resection rate, pathological resection status of patients treated with these regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proof of colorectal adenocarcinoma;
2. Age ≥ 18 years and ≤75 years;
3. RAS wild type；
4. CRS≥3；
5. Simultaneous liver-limited metastases;
6. At least one measurable liver metastases;
7. World Health Organization (WHO) performance status 0-1;
8. Life expectancy ≥ 3 months;
9. Adequate hematologic function: absolute neutrophil count (ANC)≥1.5×109/l, platelets≥100×109/l, and hemoglobin(HB) ≥ 9g/dl;
10. Adequate liver and renal function: total bilirubin ≤2.0 mg/dl, serum transaminases ≤ 5x upper limit of normal(ULN), and serum creatinine ≤ 1.5x ULN and creatinine clearance ≥ 30 ml/min;
11. Written informed consent.

Exclusion Criteria:

1. Previous systemic treatment for metastatic disease;
2. Previous surgery for metastatic disease;
3. Extrahepatic metastases;
4. Unresectable primary tumor;
5. Major cardiovascular events (myocardial infarction, severe/unstable angina, congestive heart failure, CVA) within 12 months before randomisation;
6. Acute or subacute intestinal obstruction;
7. Second primary malignancy within the past 5 years;
8. Drug or alcohol abuse;
9. No legal capacity or limited legal capacity;
10. Pregnant or lactating women;
11. Uncontrolled hypertension, or unsatisfactory blood pressure control with ≥3 antihypertensive drugs;
12. Peripheral neuropathy;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years
  The Event-free survival (EFS) was defined as the period from the start of initial medication to the date of tumor relapse, progression, or death

SECONDARY OUTCOMES:
overall survival | 5 years
  The overall survival (OS) was defined as the period from the start of initial medication until death from any cause, at which point the data was censored.
postoperative hospital stay | 30 days post operatively
  The postoperative hospital stay is defined as the number of date from the first day after operation to discharge.
postoperative complication | After surgery during one month
  Patients will be evaluated for surgical morbidity during 1 month. Postoperative morbidity will be scored according 'Clavien-Dindo Grade'.
postoperative mortality | After surgery during 90 days
  any death occured within 90 days after the last resection of primary and metastatic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hosptial, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No